CLINICAL TRIAL: NCT03578822
Title: A Phase III Trial to Assess the Efficacy and Safety of Recombinant Human Prourokinase in the Treatment of Acute Acute Ischaemic Stroke in 4.5-6 Hours After Stroke Onset
Brief Title: Thrombolysis With rhPro-UK in 4.5-6 Hours After Acute Ischemic Stroke in a Double-blinded,Controlled Trial
Acronym: PROUD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASLY-B1440-CTP-Ⅲb
Record Dates: First submitted 2018-06-20; First posted 2018-07-06 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Acute Ischaemic Stroke
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Recombinant human urokinase(rhPro-UK) and Aspirin simulation agent
  Interventions: Drug: Recombinant human urokinase; Drug: Aspirin simulation agent
- Group B (Other): rhPro-UK simulation agent and Aspirn
  Interventions: Drug: Aspirin; Drug: rhPro-UK simulation agent

INTERVENTIONS:
Drug: Recombinant human urokinase — Patients receive rhPro-UK 35mg,15mg of which is given as a bolus within 3min followed by dlivery of the remaining 20 mg as a constant infusion over a period of 30 min.
  Other Names: rhPro-UK
  Arms: Group A
Drug: Aspirin — Aspirin 300mg is taken orally at the beginning of thrombolysis.
  Arms: Group B
Drug: rhPro-UK simulation agent — Patients receive rhPro-UK simulation agent 35mg,15mg of which is given as a bolus within 3min followed by dlivery of the remaining 20 mg as a constant infusion over a period of 30 min.
  Arms: Group B
Drug: Aspirin simulation agent — Aspirin simulation agent 300mg is taken orally at the beginning of thrombolysis.
  Arms: Group A

SUMMARY:
This is a randomized,controlled, double-blinded, phase 3 clinical study to evaluate the efficacy and safety of recombinant human urokinase(rhPro-UK) versus basic treatment for patients with acute ischaemic stroke in 4.5-6 hours after stroke onset.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke with symptoms of neurological deficits.
2. Aged 18 to 80 years,male or famale.
3. NIH Stroke Scale（NIHSS）scores of 4 to 25.
4. Treatment 4.5 to 6 hours after stroke onset.(Stroke onset time is defined as the last time a patient with no clinical neurological deficit,for patients who wake up with stroke symptoms, consider that stroke occurs when the patient begins to fall asleep).
5. The symptoms of stroke last at least 30 minutes without significant improvement before treatment.
6. CT showed negative or signs of early infarction.
7. Patients and/or their families are willing to participate in this study and agree to sign informed consent.

Exclusion Criteria:

1. Patients with premorbid modified Rankin Scale(mRS) score ≥2
2. CT showed multiple infarctions（low density> 1/3 cerebral hemisphere）.
3. Transient ischemic attack.
4. Epileptic seizure when stroke onset.
5. Intracranial tumor, arteriovenous malformation and aneurysm.
6. Iatrogenic Stroke.
7. Thrombectomy is planned.
8. Cardioembolism and atrial fibrillation.
9. Myocardial infarction history within 3 months.
10. Severe cerebral trauma or stroke history within 3 months.
11. Blood pressure is still out of control after aggressive antihypertensive treatment.Uncontrolled blood pressure is defined as systolic blood pressure≥ 180mmHg or diastolic blood pressure≥100mmHg.
12. High density lesions (bleeding) and subarachnoid hemorrhage is revealed by emergency CT examination.
13. Active visceral hemorrhage.
14. Patients with intracerebral hemorrhage history.
15. Patients with diabetic retinopathy history.
16. Puncture in 1 week which can not be oppressed.
17. Major surgery or severe trauma within 2 weeks.
18. Intracranial surgery, intraspinal surgery or solid organ biopsy within 30 days.
19. Heparin treatment within 48 hours (APTT above normal upper limit).
20. Taking anticoagulant drugs orally, and PT >15s or INR >1.7.
21. High risk of acute hemorrhage include platelet count<10^9/L.
22. Taking thrombin inhibitors or factor Xa inhibitor with abnormal results of sensitive laboratory examination(e.g. APTT, INR, PLT, FIB、TT or appropriate Ⅹ a factor activity test, etc.).
23. Blood glucose < 2.7 mmol/L or > 22.2 mmol/L.
24. Pregnancy, lactating or menstrual women.
25. Patients who have difficulty swallowing and are unable to take medications orally.
26. Clinician thinks patient doesn't fit to participate in the test of other diseases or conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Functional handicap | 90days
  Proportion of patients achieving a Modified Rankin Scale(mRS,which has a range of 0 to 6, with 0 indicating no symptoms at all and 6 indicating death) of 0 to 1 at 90 days after treatment.

SECONDARY OUTCOMES:
Proportion of Neurological Improvement | 90 days
  Proportion of patients achieving a NIHSS(national institutes of health stroke scale) ≦1 or reduction of ≥4 NIHSS points at 24 hours after treatment.
Scores of Neurological Improvement | 24 hours
  NIHSS changes from baseline at 24 hours after treatment
Index Long-term Change from Baseline of Barthel Index | 90 days
  Barthel Index(which assesses the ability to perform activities of daily living, on a scale that ranges from 0 to 100) changes from baseline on 90 days after treatment.
Long-term Change from Baseline of NIHSS | 90 days
  NIHSS changes from baseline on 90 days after treatment.
Long-term Change from Baseline of mRS | 90 days
  mRS changes from baseline on 90 days after treatment.
Proportion of Long-term Improvement | 90 days
  Proportion of patients achieving a mRS of 0 to 2 at 90 days after treatment.
Proportion of Long-term Improvement | 90 days
  Proportion of patients achieving a Barthel Index of 75 to 100 at 90 days after treatment.
Systemic hemorrhage | 90days
  Severe systemic hemorrhage
Symptomatic intracerebral hemorrhage | 90days
  Symptomatic intracerebral hemorrhage (sICH)
Death | 7 days and 90 days
  Death
Recurrence | 7 days
  Recurrence of stroke

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - XuanWu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Harrison International Peace Hospital, Hengshui, Hebei
  - Tangshan Gongren Hospital, Tangshan, Hebei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Inner Mongolia People's Hospital, Hohhot, Inner Mongolia
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - The Second People'Hospital of Huai'an, Huai'an, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Pingxiang People's Hospital, Pingxiang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - Meihekou Central Hospital, Meihekou, Jilin
  - Dalian Municipal Central Hospital, Dalian, Liaoning
  - Shenyang Military Region General Hospital, Shenyang, Liaoning
  - The First People's Hospital of Shenyang, Shenyang, Liaoning
  - Luoyang Central Hospital, Luoyang, Zhengzhou